CLINICAL TRIAL: NCT05989555
Title: Effects on the Systemic Innate Immune System by Radioactive Iodine Treatment in Non-medullary Thyroid Cancer Patients
Brief Title: Effects of Radioactive Iodine on the Immune System in Thyroid Cancer
Acronym: SCIMITAR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-16623
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Thyroid Carcinoma, Nonmedullary
Keywords: radioactive iodine; innate immune system; monocytes
MeSH Terms: conditions — Thyroid Cancer, Papillary | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood mononuclear cells and monocytes will be isolated from whole blood.
  The monocytes will be stimulated in vitro. Supernatants will be stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- I/adjuvant: 15 patients with thyroid carcinoma that are treated with radioacitive iodine in an adjuvant setting
  Interventions: Other: Blood drawing
- II/structutral disease: 15 patients with thyroid carcinoma that are treated with radioactive iodine with the indication of persistent structural disease
  Interventions: Other: Blood drawing

INTERVENTIONS:
Other: Blood drawing — Blood is drawn twice in all subjects. Once before treatment with radioacitve iodine and once after.

SUMMARY:
Blood will be drawn 1 month before and 2 month after regular radioactive iodine treatment. Monocytes will be isolated. The three main outcomes are whole blood counts, cytokine production upon in vitro stimulation of monocytes and in vitro ROS production by monocytes. These results are compared between patients treated in adjuvant setting and patients treated for persistent structural disease, and between pre- and post-treatment status.

DETAILED DESCRIPTION:
Earlier studies have shown that, particularly advanced, thyroid carcinomas are highly immunogenic tumors. The immune system is involved in both pathogenesis and progression of thyroid carcinoma (TC), as in other malignancies. For example, it is known that increased tumor infiltration with tumor-associated macrophages is associated with decreased survival in TC patients. In a previous study from our group, changes in the programming of myeloid immune cells were identified in newly diagnoses TC patients. That study showed that upon stimulation, cytokine production was decreased in monocytes from TC patients when compared to monocytes from healthy volunteers or from patients with benign thyroid tumors. Also, reactive oxygen species (ROS) production (known to be tumorigenic) from monocytes was increased in TC patients when compared to healthy volunteers. In the mentioned study, several effects of radioactive iodine (RAI)-treatment, after surgery, on the systemic immune system were observed. For instance, lymphocyte counts were significantly reduced after treatment with RAI, an effect also observed in other studies. Moreover, after RAI-treatment, ROS levels produced by monocytes decreased to levels similar to those produced by monocytes of healthy controls. Although, the effect of RAI-treatment on ROS-production was less pronounced than that of surgery. There was no clear effect of RAI-treatment on the cytokine production capacity. However, it should be noted that in most patients in this study RAI was administered in a setting of remnant ablation, meaning that only a low dose of RAI was administered and that only a very low amount (or none) of cancer cells were present at the time of administration. Furthermore, the number of included patients was too low to perform subgroup analyses. The current study aims to assess the effect of RAI-treatment in patients with structural disease, as a higher dose of beta-radiation will be present in these patients, and compare these effects to that in patients treated with RAI in an adjuvant setting.

The investigators hypothesize that RAI-treatment will have a more pronounced effect on the systemic innate immune system in patients with structural disease when compared to patients treated in an adjuvant setting. This study will give us more insights in the interplay between RAI and the immune system in patients with TC.

The aim of the study is to assess the effect of RAI-treatment on the innate immune system in TC patients and to compare these effects between patients with and without structural disease in a prospective explorative study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed non-medullary thyroid cancer
* Undergoing radioactive iodine treatment in an adjuvant setting or for persistent structural disease
* Aged ≥ 18 years

Exclusion Criteria:

* Inflammatory or infectious comorbidities
* Using medication interfering with the immune system
* Pregnancy
* A self-reported alcohol consumption of >21 units per week
* Other active malignancies, defined as malignancies not in complete remission for <2 years
* Previous systemic anti-cancer treatment such as chemotherapy, targeted therapy, radiotherapy or immunotherapy within 3 years before study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty patients with non-medulary thyroid carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Whole blood counts | 2 months
  Whole blood counts with leukocyte subtypes (neutrophils, lymphocytes and monocytes) are compared before and after radioactive iodine treatment
Cytokine production upon monocyte stimulation | 2 months
  Cytokine produciton (tumor necrosis factor, interleukin-6, interleukin-8) will be compared before and after treatment with radioactive iodine
Reactive oxygen species (ROS) production by monocytes | 2 months
  In vitro ROS production by monocytes will be compared before and after treatment with radioactive iodine

SECONDARY OUTCOMES:
Monocyte transcriptome | 2 months
  Possibly, transcriptome of monocytes will be compared before and after treatment with radioactive iodine
Plasma proteome | 2 months
  Possibly, plasma proteome (especially inflammatory markers) will be compared before and treatment with radioactive iodine.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided